CLINICAL TRIAL: NCT03323684
Title: Analgesic Efficacy of Ultrasound-guided Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Laparoscopic Cholecystectomy
Brief Title: Quadratus Lumborum Block vs Transversus Abdominis Plane Block for Post-cholecystectomy Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MD/17.09.09
Record Dates: First submitted 2017-10-17; First posted 2017-10-27 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Control Groups; Fentanyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadratus lumborum block Group (QL) (Experimental): Quadratus lumborum block will be performed
  Interventions: Other: Quadratus lumborum block Group (QL); Drug: Paracetamol infusion; Drug: Ketorolac analgesia; Drug: fentanyl
- Transversus abdominis plane Group (TAP) (Experimental): Subcostal transversus abdominis plane will be performed
  Interventions: Other: Transversus abdominis plane Group (TAP); Drug: Paracetamol infusion; Drug: Ketorolac analgesia; Drug: fentanyl
- Control group (C) (Experimental): Postoperative analgesia will be accomplished with conjunction of paracetamol and ketorolac
  Interventions: Other: Control group (C); Drug: Paracetamol infusion; Drug: Ketorolac analgesia; Drug: fentanyl

INTERVENTIONS:
Other: Quadratus lumborum block Group (QL) — 20 mL of 0.375% isobaric bupivacaine for each side deposited at the posterior aspect of the quadratus lumborum muscle (QLB type 2) using ultrasound after induction of general anesthesia and 15 minutes before start of surgery
  Arms: Quadratus lumborum block Group (QL)
Other: Transversus abdominis plane Group (TAP) — 20 mL of 0.375% isobaric bupivacaine for each side using ultrasound after induction of general anesthesia and 15 minutes before start of surgery
  Arms: Transversus abdominis plane Group (TAP)
Other: Control group (C) — No intervention will be done
  Arms: Control group (C)
Drug: Paracetamol infusion — Paracetamol infusion (15 mg.kg) will be given by intravenous infusion after induction of general anesthesia.
Drug: Ketorolac analgesia — In PACU Ketorolac 30 mg ampoule will be given by intravenous infusion to all cases and then every 8 hours.
Drug: fentanyl — With induction of general anaesthesia, fentanyl (1 microgram.kg) will be given. Intraoperatively, Fentanyl boluses (0.5 microgram.kg) will be given in case of increase in intraoperative mean arterial blood pressure or heart rate of more than 20% of baseline for longer than 5 minutes. Postoperatively, Fentanyl boluses (20 micrograms) will be given if VAS is more than 3 and it might be repeated after 30 minutes until VAS is ≤ 3.

SUMMARY:
In laparoscopic cholecystectomy, overall pain is a conglomerate of three different and clinically separate components: incisional pain (somatic pain) due to trocar insertion sites, visceral pain (deep intra abdominal pain), and shoulder pain due to peritoneal stretching and diaphragmatic irritation associated with carbon dioxide insufflation. Moreover, it has been hypothesized that intense acute pain after laparoscopic cholecystectomy may predict development of chronic pain (e.g., postlaparoscopic cholecystectomy syndrome). Without effective treatment, this ongoing pain may delay recovery, mandate inpatient admission, and thereby increase the cost of such care.

Recently, the uses of peripheral axial blocks that deliver local anesthetic into the transversus abdominis fascial plane have become popular for operations that involve incision(s) of the abdominal wall. Thus, the Transversus Abdominis plane (TAP) block has been shown to reduce perioperative opioid use in elective abdominal surgery, including open appendicectomy, laparotomy, and laparoscopic cholecystectomy. However, the efficacy of the TAP block is reportedly only reliable in providing analgesia below the umbilicus. The ultrasound-guided subcostal transversus abdominis (STA) block is a recently described variation on the TAP block which produces reliable supraumbilical analgesia. Deposition of local anesthetic in this plane has shown to block dermatomes T6 to T10 with an occasional spread to T12. This variant will be discussed in our study.

Currently, the Quadratus Lumborum block (QL block) is performed as one of the perioperative pain management procedures for all generations (pediatrics, pregnant, and adult) undergoing abdominal surgery. The local anesthetic injected via the approach of the posterior QL block ( QL 2 block ) can more easily extend beyond the TAP to the thoracic paravertebral space or the thoracolumbar plane, the posterior QL block entails a broader sensory-level analgesic and may generate analgesia from T7 to L1. Use of posterior QL block in laparoscopic cholecystectomy has not been investigated before and it is the variant that will be discussed in our study.

DETAILED DESCRIPTION:
The aim of this study is to compare the analgesic efficacy of ultrasound guided posterior quadratus lumborum block and subcostal transversus abdominis plane block in laparoscopic cholecystectomy. The primary outcome will be assessment of postoperative opioid analgesic requirements. The secondary outcomes will include assessing intraoperative analgesic requirements, stress of trocar insertion and insufflation, postoperative visual analogue scale (VAS), length of stay at post-anesthesia care unit (PACU), time of first request to analgesia, incidence of nausea, and vomiting.

The study will hypothesize that quadratus lumborum block will be more superior than or equal to transversus abdominis block because it could cover all the dermatome segments from caudally L1 to cranially till T6 segments as the drug is expected to travel from the QL to the higher paravertebral spaces.

ELIGIBILITY:
Inclusion Criteria:

* American Physical Status I or II

Exclusion Criteria:

* Patient refusal.
* Hematological diseases
* bleeding disorders.
* Coagulation abnormality.
* Psychiatric diseases.
* Local skin infection
* sepsis at site of the block.
* Known intolerance to the study drugs.
* Body Mass Index > 40 Kg/m2.
* Emergency laparoscopic cholecystectomy
* if laparoscopic procedure converted to open.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Cumulative postoperative fentanyl consumption (total dose given in micrograms) | For 24 hours after surgery

SECONDARY OUTCOMES:
Cumulative intraoperative fentanyl consumption (total dose given in micrograms) | For 4 hours after start of anaesthesia
  Cumulative use of fentanyl during intra-operative period
Heart rate | For 4 hours after start of anaesthesia
  Changes in intra-operative heart rate values
Mean arterial blood pressure (mmHg) | For 4 hours after start of anaesthesia
  Changes in intra-operative mean arterial blood pressure values
Dermatomal distribution of the extent of the blockade will be assessed by pinprick method | the first one hour after surgery
  Assessment of dermatomal distribution of the block for evaluating the success or failure of the block
Postoperative pain severity will be assessed using VAS | For 24 hours after surgery
  The severity of postoperative pain will be measured and recorded by using the visual analogue scale (VAS) for pain, where 0 is equal to no pain and 10 indicates the worst possible pain
Time for the first request to rescue analgesia (in minutes) | For 24 hours after surgery
  Time for first request to rescue analgesia
length of stay at PACU (in minutes) | For 24 hours after surgery
Incidence of postoperative nausea and vomiting | For 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Y Makharita, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care
Locations (2):
- Egypt (2):
  - Mansoura University, Faculty of Medicine, Al Mansurah, DK
  - Mansoura University, Al Mansurah, DK

IPD SHARING:
Plan to Share IPD: Undecided